CLINICAL TRIAL: NCT07351773
Title: Autonomic Neuromodulation With Ultrasound-Guided Stellate Ganglion Block in Alzheimer's Disease: A Randomized Controlled Trial
Brief Title: Ultrasound-Guided Stellate Ganglion Block for Alzheimer's Disease
Acronym: SGB-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taizhou Second People's Hospital (Other)
Collaborators: Taizhou Municipal Bureau of Science and Technology (Unknown)
Responsible Party: Principal Investigator, Yanan Ge, Attending Physician, Taizhou Second People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TZYE-KY-2024-003; 24ywb104 (Other Grant/Funding Number: Taizhou Municipal Science and Technology Bureau)
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease(AD); Cognitive Dysfunction
Keywords: Stellate Ganglion Block; Ultrasound-Guided; Autonomic Nervous System; Cognition; Mini-Mental State Examination; Randomized Controlled Trial; Quality of Life; Anxiety; Depression; Instrumental Activities of Daily Living
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Anxiety Disorders; Depression | interventions — Memantine; Donepezil

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group trial comparing ultrasound-guided stellate ganglion block plus standard drug treatment versus standard drug treatment alone.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-Guided SGB Plus Standard Drug Treatment (Experimental): Participants receive ultrasound-guided stellate ganglion block (SGB) in addition to standard-of-care Alzheimer's pharmacotherapy (memantine and/or donepezil) based on pre-existing treatment history; not all participants receive both medications.
  Interventions: Procedure: Ultrasound-Guided Stellate Ganglion Block; Drug: Memantine hydrochloride; Drug: Donepezil hydrochloride
- Standard Drug Treatment Alone (Active Comparator): Participants receive standard drug treatment alone without stellate ganglion block. Participants received standard-of-care Alzheimer's pharmacotherapy (memantine and/or donepezil) based on pre-existing treatment history; not all participants received both medications.
  Interventions: Drug: Memantine hydrochloride; Drug: Donepezil hydrochloride

INTERVENTIONS:
Procedure: Ultrasound-Guided Stellate Ganglion Block — Ultrasound-guided stellate ganglion block performed according to a standardized protocol. The procedure was administered as a treatment course consisting of 10 sessions on alternate days.
  Other Names: SGB
  Arms: Ultrasound-Guided SGB Plus Standard Drug Treatment
Drug: Memantine hydrochloride — Background standard-of-care pharmacotherapy for Alzheimer's disease. Participants continued their pre-enrollment memantine regimen as clinically indicated. Treatment could include memantine alone or in combination with donepezil. Dose and schedule were not standardized and were determined by the treating physician based on prior treatment history and routine clinical practice; all medication use and any changes were recorded.
Drug: Donepezil hydrochloride — Background standard-of-care pharmacotherapy for Alzheimer's disease. Participants continued their pre-enrollment donepezil regimen as clinically indicated. Treatment could include donepezil alone or in combination with memantine. Dose and schedule were not standardized and were determined by the treating physician based on prior treatment history and routine clinical practice; all medication use and any changes were recorded.

SUMMARY:
The goal of this clinical trial is to learn if ultrasound-guided stellate ganglion block (SGB), added to standard drug treatment, can improve thinking and memory in people with Alzheimer's disease. It will also learn about the safety of SGB.

The main questions this study aims to answer are:

Do people who receive SGB plus standard drug treatment have better global cognition, measured by the Mini-Mental State Examination (MMSE), 1 month after finishing the treatment course compared with people who receive standard drug treatment alone? How do anxiety, depression, quality of life, and ability to live independently change over 1 month, 3 months, and 6 months after treatment? What medical problems, if any, occur during or after SGB?

Researchers will compare two groups:

SGB plus standard drug treatment Standard drug treatment alone

Participants will:

Be randomly assigned to one of the two groups Receive the assigned treatment Complete study visits and assessments at baseline and at 1 month, 3 months, and 6 months after finishing the treatment course

DETAILED DESCRIPTION:
This is a randomized, parallel-group clinical trial in people with Alzheimer's disease. Participants are assigned to receive either ultrasound-guided stellate ganglion block (SGB) in addition to standard drug treatment or standard drug treatment alone. SGB is a procedure performed under ultrasound guidance in the neck region to temporarily block the stellate ganglion, which may influence autonomic nervous system activity.

The primary outcome is global cognition measured by the Mini-Mental State Examination (MMSE). The prespecified primary endpoint is 1 month after completion of the treatment course to capture a relatively stable post-treatment effect. Secondary outcomes include anxiety symptoms measured by the Zung Self-Rating Anxiety Scale (SAS), depressive symptoms measured by the Zung Self-Rating Depression Scale (SDS), quality of life measured by the Alzheimer's Disease Quality of Life scale (QoL-AD), and independent living ability measured by the Lawton-Brody Instrumental Activities of Daily Living scale (IADL). Outcomes are assessed at baseline and at 1 month, 3 months, and 6 months after completion of the treatment course.

Safety is evaluated by monitoring and recording adverse events related to the procedure and study participation throughout the treatment period and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 to 85 years.
2. Diagnosis of Alzheimer's disease (AD) based on the 2011 NIA-AA criteria.
3. Mild to moderate cognitive impairment assessed by the Mini-Mental State Examination (MMSE).
4. Ability to understand study procedures and provide written informed consent by the participant or a legally authorized representative.
5. Ability to complete scheduled follow-up assessments.

Exclusion Criteria:

1. Known allergy to lidocaine, coagulation disorders, or other contraindications to stellate ganglion block (SGB).
2. Severe cardiac, hepatic, or renal disease that could compromise safety.
3. Cranial surgery or major head trauma within the past 6 months.
4. Participation in other interventional trials that could affect study outcomes.
5. Cognitive impairment primarily due to other neurodegenerative diseases or psychiatric disorders.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-26 (Actual); Primary Completion 2025-06-29 (Actual); Study Completion 2025-11-29 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) Total Score | Baseline; Day 20 (end of treatment course); and 1, 3, and 6 months after completion of the treatment course.
  Global cognition assessed using the Mini-Mental State Examination (MMSE). Total score range 0-30; higher scores indicate better cognitive function. The prespecified primary endpoint is 1 month after completion of the treatment course.

SECONDARY OUTCOMES:
Zung Self-Rating Anxiety Scale (SAS) Standard Score | Baseline; Day 20 (end of treatment course); and 1, 3, and 6 months after treatment completion.
  Anxiety symptoms assessed using the Zung Self-Rating Anxiety Scale (SAS). The raw total score is multiplied by 1.25 and rounded to obtain a standard score. Score range 25-100; higher scores indicate more severe anxiety.
Zung Self-Rating Depression Scale (SDS) Standard Score | Baseline; Day 20 (end of treatment course); and 1, 3, and 6 months after treatment completion.
  Depressive symptoms assessed using the Zung Self-Rating Depression Scale (SDS). The raw total score is multiplied by 1.25 and rounded to obtain a standard score. Score range 25-100; higher scores indicate more severe depressive symptoms.
Quality of Life in Alzheimer's Disease (QoL-AD) Total Score | Baseline; Day 20 (end of treatment course); and 1, 3, and 6 months after treatment completion.
  Quality of life assessed using the Quality of Life in Alzheimer's Disease scale (QoL-AD). Total score range 13-52; higher scores indicate better quality of life.
Lawton-Brody Instrumental Activities of Daily Living (IADL) Total Score | Baseline; Day 20 (end of treatment course); and 1, 3, and 6 months after treatment completion.
  Independent living ability assessed using the Lawton-Brody Instrumental Activities of Daily Living scale (IADL). Total score range 8-24; lower scores indicate poorer independence and greater care needs.
Procedure-Related Adverse Events | Periprocedural (Day 1 through Day 20): during each stellate ganglion block session and within 30 minutes after each session.
  Number of participants with procedure-related adverse events occurring during the stellate ganglion block procedure or within 30 minutes after each session.

CONTACTS AND LOCATIONS:
Overall Officials: Yanan Ge, Principal Investigator — Taizhou Second People's Hospital
Locations (1):
- Taizhou Second People's Hospital, Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive clinical information, and public or external sharing is not permitted under the informed consent, ethics approval requirements, and institutional policies. To protect participant privacy and confidentiality, only aggregated, de-identified results will be reported.